CLINICAL TRIAL: NCT05345431
Title: Endovascular Denervation for the Treatment of Patients With Peripheral Arterial Disease
Acronym: EDPAD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Zhongda Hospital (Other)
Responsible Party: Principal Investigator, Gao-jun Teng, Clinical Professor, Zhongda Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EDN-PAD
Record Dates: First submitted 2022-04-12; First posted 2022-04-25 (Actual); Last update posted 2022-04-25 (Actual); Status verified 2022-04

CONDITIONS: PAD

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The control group (Other): Treating with balloon dilation or stent implantation only,
  Interventions: Device: PTA
- The EDN group (Experimental): Treating with EDN at the site of the iliac artery distal to the superficial femoral artery proximal before balloon dilation or stent implantation.
  Interventions: Device: endovascular denervation

INTERVENTIONS:
Device: endovascular denervation — Treating with EDN at the site of the iliac artery distal to the superficial femoral artery proximal before balloon dilation or stent implantation
  Arms: The EDN group
Device: PTA — Treating with balloon dilation or stent implantation
  Arms: The control group

SUMMARY:
Sympathetic overactivity partly promotes the development of peripheral artery disease which mainly leads to ischemia of the lower limbs. Endovascular arterial denervation (ED) is a minimally invasive technique which could deliver Radiofrequency energy by a multi-electrode catheter to the Lower limb artery to restore Sympathetic activity. The purpose of this study is to evaluate the effects of multi-electrode radiofrequency ablation system on lower limb ischemia with PAD.

DETAILED DESCRIPTION:
Peripheral arterial disease(PAD) show insufficient blood supply of diseased limbs, which causes intermittent claudication of lower limbs, reduced skin temperature, pain, and chronic progressive disease that still produces ulcer or necrosis. Some clinical studies have shown Sympathetic overactivity in the lower arterial ischemic disease. The multi-electrode radiofrequency ablation system can significantly reduce the excitability of sympathetic nerve, restore the normal response of sympathetic nerve, relieve the pain and discomfort of patients, effectively improve the symptoms of lower limb ischemia, and improve the quality of life of patients.

ELIGIBILITY:
Inclusion Criteria:

1. eligible subjects aged 18-75 years,
2. clinically confirmed PAD patients in Rutherford category II-VI.

Exclusion Criteria:

1. thrombolytic therapy performed within 30 days,
2. patients who had undergone vascular bypass surgery before this study,
3. allergy or contraindication of antiplatelet drugs, anticoagulants, thrombolytic drugs and contrast agents,
4. patients with obvious bleeding tendency, coagulation dysfunction, hypercoagulability and blood system diseases,
5. serious liver and kidney diseases,
6. history of hemorrhagic stroke within the last 1 month or ischemic stroke or transient ischemic attack within 2 weeks,
7. pacemaker implants,
8. patients who are pregnant, breast-feeding or planning pregnancy,
9. expected survival < 24 months.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2022-04-25 (Estimated); Primary Completion 2025-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Ischemia relief | from baseline to 6 months after procedure
  Changes of the ankle brachial index(ABI)

SECONDARY OUTCOMES:
Ischemia relief | from baseline to 3 months after procedure
  Changes of the ankle brachial index(ABI)
clinical benefit | from baseline to 3, 6 months after procedure
  Changes of the Rutherford category(Rutherford category includes a total of 0-6 grades, the lower the grade, the better the results)
pain relief | from baseline to 3 ,6 months after procedure
  Changes of the numeric rating scale ( NRS) scores(NRS scores includes a total of 0-10 grades, the lower the grade, the better the results)

CONTACTS AND LOCATIONS:
Overall Officials: Gao-Jun Teng, MD, Principal Investigator — Zhongda Hospital
Locations (1):
- Zhongda Hospital, Southeast University, Nanjing, Jiangsu, China